CLINICAL TRIAL: NCT01836744
Title: Survival Rate of Dental Implants Placed in Sinus Lift Performed With Two Different Grafts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grupo de Investigação: Cirurgia Oral, Peridontologia, Implantologia (Other)
Collaborators: Universidade do Porto (Other); Dentsply Sirona Implants and Consumables (Industry); Tecnoss OsteoBiol (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D-2012-024
Record Dates: First submitted 2013-03-11; First posted 2013-04-22 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Dental Implant Survival Rate

STUDY DESIGN:
Intervention Model Description: randomizes split month trial:
  * one sinus autologous bone graft
  * other sinus - xenograft - osteobiol Mp3
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Seal envelops, codification of the side and patient and independent blind assessors
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- survival rate autologous bone (Active Comparator): dental implant placement in the previous sinus lift side with autologous bone; dental implant placement in the previous sinus lift side with xenograft material side;
  Interventions: Device: Survival rate dental implant (OsseoSpeed™)
- survival rate axenograft material (Active Comparator): dental implant placement in the previous sinus lift side with xenograft material side;
  Interventions: Device: Survival rate dental implant (OsseoSpeed™)

INTERVENTIONS:
Device: Survival rate dental implant (OsseoSpeed™)
  Other Names: OsseoSpeed™ dental implant

SUMMARY:
Previous in a randomized way, it will be performance 12 bilateral sinus lift with autologous bone in one side and the in other with xenograft material. After 6 mouths we will place 1 to 3 implants in each side and analyse the survival rate and possibles differences related to; prosthesis failure; biological and prosthetic complications; peri-implant marginal bone level changes.

DETAILED DESCRIPTION:
The study will be performance in 12 patients submitted to a bilateral sinus lift procedure.

Six months after the bilateral sinus lifting performed in a randomly way, using as graft materials (100% of autologous bone graft or 100% of xenograft), will be placed 1 to 3 implants in each maxillary sinus.

Wait more six months to expose the implant. At the end of 13 months after implant placement it should be in charge.

Implant placement (6 months after sinus lift procedure):

* Both sides should be treated during the same session.
* Patients will receive 2g Amoxicillin one hour before the procedure. Patients allergic to penicillin will be given Clindamycin 600 mg 1 hour before implant placement procedure.
* Patients will rinse for 1 minute prior to flap elevation with 0.12% chlorhexidine mouthwash.
* After delivery of local anaesthesia, incision and flap elevation, the recommendation of the various implant manufacturers will be followed for placing 1 to 3 implants 9-11 mm long per posterior upper (premolar-molar areas) below the maxillary sinus and a histological sample for each side will be collected.
* The neck of the implants will be placed flush to the bone and implants will be submerged under the soft tissues and flaps will be sutured.
* Baseline intraoral radiographs of the study implants have to be taken.

Post-implant placement instructions:

* Chlorhexidine mouthwash 0.12% for 1 minute twice a day for 2 weeks.
* Ibuprofen 400 mg will be prescribed to be taken 2-4 times a day during meals, but patients will be instructed not to take them in absence of pain. Patients with gastric problems or allergic to ibuprofen will receive paracetamol 1 g instead.
* Sutures will be removed after 10 days.

Abutment connection (6 months after implant placement):

* Both sides should be treated during the same session.
* Patients will rinse for 1 minute prior to flap incision with 0.12% chlorhexidine mouthwash.
* Mucosa can be punched or a flap will be elevated according to personal preference of the surgeon, it is important that both sides are treated in the same way.
* Individual implants will be tested for stability.
* Impressions will be taken.
* Healing abutments will be placed.

Post-abutment connection instructions:

* Chlorhexidine mouthwash 0.12% for 1 minute twice a day for 2 weeks.
* Ibuprofen 400 mg will be prescribed to be taken 2-4 times a day during meals, but patients will be instructed not to take them in absence of pain. Patients with gastric problems or allergic to ibuprofen will receive paracetamol 1 g instead.
* Sutures will be removed after 10 days.

Prosthetic phase:

* Within one month after abutment connection, implants will be manually tested for stability.
* Provisional reinforced acrylic restorations or definitive screw-retained or provisionally cemented (to allow implant stability assessment) metal-resin or metal-ceramic bridges rigidly joining the 2 or 3 implants will be delivered.
* Implants will be splinted under the same prosthesis, each implant supporting one tooth element.
* The connection of teeth with implants under the same prosthesis is not allowed.
* Similar procedures and materials have to be used in the same patient.
* The occlusal surface will be in slight contact with the opposite dentition.
* Intraoral radiographs and clinical pictures of the study implants will be taken at initial loading.

Maintenance:

* All patients will be recalled every 6 months after prosthetic loading for delivery of professional maintenance on individual basis.
* Dental occlusion will be evaluated at each maintenance visit.

ELIGIBILITY:
Inclusion Criteria:

* Any partially edentulous patient having bilateral edentulism in the posterior maxillae (premolars and/or molars) with a similar degree of bone resorption requiring one to three implants at each side, being 18 years or older, and able to sign an informed consent. For all the potentially included patients preoperative CBCT (cone beam computed tomography) or CT scans and OPGs (orthopantomograph)must be obtained and attached to the files. The vertical bone height below the maxillary sinus at the implant sites must be of 1-5 mm and bone thickness at least 6 mm measured on CBCT (cone-beam computed tomography)or CT scans. Smokers will be included and patients will be grouped into: 1) non smokers; 2) light smokers ≤ 10 cigarettes/day; 3) heavy smokers ≥ 11 cigarettes/day, according to what they declare.

Exclusion Criteria:

* General contraindications to implant surgery.
* Patients irradiated in the head and neck area.
* Immunosuppressed or immunocompromised patients.
* Patients treated or under treatment with intravenous amino-bisphosphonates.
* Patients with untreated periodontitis.
* Patients with poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnancy or nursing.
* Substance abuser.
* Psychiatric problems or unrealistic expectations.
* Lack of opposite occluding dentition in the area intended for implant placement.
* Patients with an acute or chronic sinusitis.
* Patients participating in other trials, if the present protocol cannot be properly adhered too.
* Patients referred only for implant placement.
* Patient unable to be followed for 5 years after loading.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Histological and histomorphological analysis | 6 mounths
  Histological and histomorphological analysis of the bone graft
radiological analysis | 6 mounths
  Comparation of the bone gain in a radiological analysis (initial and at 6 months)
Clinical evaluation - questionary | 6 mounths
  questionary about patient preference treatment
Implant failure | up to 5 years of loading
  implant mobility assessed manually with the removed prosthesis and/or any infection dictating implant removal. Assessments will be done at delivery of the provisional and definitive prostheses, 1, 3 and 5 years of loading by tightening the abutment screws with the removed prostheses.
Prosthesis failure | up to 5 years of loading
  when prosthesis placement will not be possible due to implant failure or secondary to implant failure.
Peri-implant marginal bone level changes | up to 5 years
  Peri-implant marginal bone level changes assessed on periapical radiographs taken with the paralleling technique at implant placement, at initial prosthetic loading, 1 and 5 years follow-up in function.
  The distance between marginal bone level and implant/abutment junction, approximated to half mm, will be measured at both mesial and distal sides and averaged. Bone level changes at single implants will be averaged at patients level and then at group level.
Biological complications | up to 5 years
  Biological complications (number and type). Particular attention will be used to assess possible sinus pathologies.
Prosthetic complications | up to 5 years
  Prosthetic complications (number and type).

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Correia, DDS, Msc, PhD, Principal Investigator — Universidade do Porto; Ricardo Faria Almeida, DDS, Msc, PhD, Study Director — Universidade do Porto; Antonio Campos Felino, DDS, PhD, Study Chair — Universidade do Porto; Sonia Gouveia, Phd, Study Chair — Instituto de Engenharia Eletrónica e Informática de Aveiro (IEETA/UA) and Centro de I&D em Matemática e Aplicações (CIDMA/UA), Universidade de Aveiro (UA), Portugal; Daniel H Pozza, DDS, PhD, Study Chair — Departamento de Biomedicina da Faculdade de Medicina, and Faculdade de Ciências da Nutrição e Alimentação, and I3s, Universidade do Porto, Porto, Portugal.
Locations (1):
- University of Porto, Faculty of Dental Medicine, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/20238367